CLINICAL TRIAL: NCT02066415
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of AMG 334 in Chronic Migraine Prevention
Brief Title: A Study to Evaluate the Efficacy and Safety of Erenumab (AMG 334) in Chronic Migraine Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20120295; 2013-001707-36 (EudraCT Number)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2018-06-21 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Treatment for Prevention of Chronic Migraine
Keywords: Chronic Migraine
MeSH Terms: interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo on day 1 and at weeks 4 and 8 by subcutaneous injection.
  Interventions: Drug: Placebo
- Erenumab 70 mg (Experimental): Participants received 70 mg erenumab on day 1 and at weeks 4 and 8 by subcutaneous injection.
  Interventions: Biological: Erenumab
- Erenumab 140 mg (Placebo Comparator): Participants received 140 mg erenumab on day 1 and at weeks 4 and 8 by subcutaneous injection.
  Interventions: Biological: Erenumab

INTERVENTIONS:
Biological: Erenumab — Administered once a month subcutaneously by authorized investigational site study staff.
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab 140 mg; Erenumab 70 mg
Drug: Placebo — Administered once a month subcutaneously by authorized investigational site study staff.
  Arms: Placebo

SUMMARY:
To evaluate the effect of erenumab compared to placebo on the change from baseline in the number of monthly migraine days in adults with chronic migraine.

DETAILED DESCRIPTION:
This study consisted of the following phases: screening, 4-week baseline phase, 12-week double-blind treatment, and 12-week follow-up. Participants may have elected to participate in the optional pharmacokinetic substudy and the optional, novel patient-reported outcome (PRO) assessment substudy.

Participants who completed the 12-week double-blind treatment phase of Study 20120295 were eligible to enroll in an open-label extension study (Study 20130255; NCT02174861).

ELIGIBILITY:
Inclusion Criteria:

* History of at least 5 attacks of migraine without aura and/or migraine with visual sensory, speech and/or language, retinal or brainstem aura.
* History of ≥ 15 headache days per month of which ≥ 8 headache days were assessed by the subject as migraine day.
* ≥ 4 distinct headache episodes, each lasting ≥ 4 hours OR if shorter, associated with use of a triptan or ergot-derivative on the same calendar day based on the eDiary calculations.
* Demonstrated at least 80% compliance with the eDiary.

Exclusion Criteria:

* History of cluster headache or hemiplegic migraine headache
* Unable to differentiate migraine from other headaches
* Failed > 3 medication categories due to lack of efficacy for prophylactic treatment of migraine .
* Received botulinum toxinin head or neck region within 4 months prior to screening.
* Used a prohibited migraine prophylactic medication, device or procedure within 2 months prior to the start of the baseline phase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2016-02-24 (Actual); Study Completion 2016-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (66):
- United States (33):
  - Research Site, La Jolla, California
  - Research Site, Newport Beach, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Sherman Oaks, California
  - Research Site, Stanford, California
  - Research Site, Stamford, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Pikesville, Maryland
  - Research Site, Watertown, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Reno, Nevada
  - Research Site, Amherst, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Temple, Texas
  - Research Site, Virginia Beach, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Montreal, Quebec
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- Research Site, Glostrup Municipality, Denmark
- Finland (5):
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Oulu
  - Research Site, Tampere
  - Research Site, Turku
- Germany (6):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Königstein im Taunus
- Norway (4):
  - Research Site, Ålesund
  - Research Site, Lillehammar
  - Research Site, Sandvika
  - Research Site, Stavanger
- Poland (6):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Świdnik
  - Research Site, Warsaw
- Sweden (3):
  - Research Site, Falköping
  - Research Site, Stockholm
  - Research Site, Vällingby
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Hull
  - Research Site, London
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Background] Tepper S, Ashina M, Reuter U, Brandes JL, Dolezil D, Silberstein S, Winner P, Leonardi D, Mikol D, Lenz R. Safety and efficacy of erenumab for preventive treatment of chronic migraine: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2017 Jun;16(6):425-434. doi: 10.1016/S1474-4422(17)30083-2. Epub 2017 Apr 28. PMID 28460892
- [Background] Cheng S, Picard H, Zhang F, Eisele O, Mikol DD. Efficacy and safety of erenumab for migraine prevention: an overview. Japanese Journal of Headache. 2019; 45 : 493-505.
- [Background] Zhou Y, Zhang F, Starcevic Manning M, Hu Z, Hsu CP, Chen PW, Peng C, Loop B, Mytych DT, Paiva da Silva Lima G. Immunogenicity of erenumab: A pooled analysis of six placebo-controlled trials with long-term extensions. Cephalalgia. 2022 Jul;42(8):749-760. doi: 10.1177/03331024221075621. Epub 2022 Mar 10. PMID 35272533
- [Background] Ashina M, Kudrow D, Reuter U, Dolezil D, Silberstein S, Tepper SJ, Xue F, Picard H, Zhang F, Wang A, Zhou Y, Hong F, Klatt J, Mikol DD. Long-term tolerability and nonvascular safety of erenumab, a novel calcitonin gene-related peptide receptor antagonist for prevention of migraine: A pooled analysis of four placebo-controlled trials with long-term extensions. Cephalalgia. 2019 Dec;39(14):1798-1808. doi: 10.1177/0333102419888222. Epub 2019 Nov 10. PMID 31707815
- [Background] Kudrow D, Pascual J, Winner PK, Dodick DW, Tepper SJ, Reuter U, Hong F, Klatt J, Zhang F, Cheng S, Picard H, Eisele O, Wang J, Latham JN, Mikol DD. Vascular safety of erenumab for migraine prevention. Neurology. 2020 Feb 4;94(5):e497-e510. doi: 10.1212/WNL.0000000000008743. Epub 2019 Dec 18. PMID 31852816
- [Background] Lipton RB, Burstein R, Buse DC, Dodick DW, Koukakis R, Klatt J, Cheng S, Chou DE. Efficacy of erenumab in chronic migraine patients with and without ictal allodynia. Cephalalgia. 2021 Oct;41(11-12):1152-1160. doi: 10.1177/03331024211010305. Epub 2021 May 13. PMID 33982623
- [Background] Lipton RB, Dodick DW, Kudrow D, Reuter U, Tenenbaum N, Zhang F, Lima GPDS, Chou DE, Mikol DD. Reduction in migraine pain intensity in patients treated with erenumab: A post hoc analysis of two pivotal randomized studies. Cephalalgia. 2021 Dec;41(14):1458-1466. doi: 10.1177/03331024211028966. Epub 2021 Aug 18. PMID 34407654
- [Background] Lipton RB, Tepper SJ, Reuter U, Silberstein S, Stewart WF, Nilsen J, Leonardi DK, Desai P, Cheng S, Mikol DD, Lenz R. Erenumab in chronic migraine: Patient-reported outcomes in a randomized double-blind study. Neurology. 2019 May 7;92(19):e2250-e2260. doi: 10.1212/WNL.0000000000007452. Epub 2019 Apr 17. PMID 30996060
- [Background] Lipton RB, Tepper SJ, Silberstein SD, Kudrow D, Ashina M, Reuter U, Dodick DW, Zhang F, Rippon GA, Cheng S, Mikol DD. Reversion from chronic migraine to episodic migraine following treatment with erenumab: Results of a post-hoc analysis of a randomized, 12-week, double-blind study and a 52-week, open-label extension. Cephalalgia. 2021 Jan;41(1):6-16. doi: 10.1177/0333102420973994. Epub 2020 Dec 3. PMID 33269951
- [Background] Tepper SJ, Diener HC, Ashina M, Brandes JL, Friedman DI, Reuter U, Cheng S, Nilsen J, Leonardi DK, Lenz RA, Mikol DD. Erenumab in chronic migraine with medication overuse: Subgroup analysis of a randomized trial. Neurology. 2019 May 14;92(20):e2309-e2320. doi: 10.1212/WNL.0000000000007497. Epub 2019 Apr 17. PMID 30996056
- [Derived] Lampl C, Kraus V, Lehner K, Loop B, Chehrenama M, Maczynska Z, Ritter S, Klatt J, Snellman J. Safety and tolerability of erenumab in individuals with episodic or chronic migraine across age groups: a pooled analysis of placebo-controlled trials. J Headache Pain. 2022 Aug 18;23(1):104. doi: 10.1186/s10194-022-01470-4. PMID 35978286
- [Derived] Ashina M, Goadsby PJ, Dodick DW, Tepper SJ, Xue F, Zhang F, Brennan F, Paiva da Silva Lima G. Assessment of Erenumab Safety and Efficacy in Patients With Migraine With and Without Aura: A Secondary Analysis of Randomized Clinical Trials. JAMA Neurol. 2022 Feb 1;79(2):159-168. doi: 10.1001/jamaneurol.2021.4678. PMID 34928306
- [Derived] Tepper SJ, Ashina M, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Picard H, Cheng S, Chou DE, Zhang F, Klatt J, Mikol DD. Reduction in acute migraine-specific and non-specific medication use in patients treated with erenumab: post-hoc analyses of episodic and chronic migraine clinical trials. J Headache Pain. 2021 Jul 23;22(1):81. doi: 10.1186/s10194-021-01292-w. PMID 34301173
- [Derived] Brandes JL, Diener HC, Dolezil D, Freeman MC, McAllister PJ, Winner P, Klatt J, Cheng S, Zhang F, Wen S, Ritter S, Lenz RA, Mikol DD. The spectrum of response to erenumab in patients with chronic migraine and subgroup analysis of patients achieving >/=50%, >/=75%, and 100% response. Cephalalgia. 2020 Jan;40(1):28-38. doi: 10.1177/0333102419894559. Epub 2019 Dec 9. PMID 31816249
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 69 centers in Canada, Czech Republic, Denmark, Germany, Finland, Norway, Poland, Sweden, United Kingdom, and the United States of America (USA).
  The first participant was enrolled on 05 March 2014 and the last participant enrolled on 05 November 2015.
Pre-assignment Details: Participants were randomized in a 3:2:2 ratio to receive placebo, erenumab 70 mg, or erenumab 140 mg. Randomization was stratified by region (North America vs Other) and medication overuse status at baseline (Yes vs No).
Period: Overall Study
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg
Started | 286 | 191 | 190
Received Study Drug | 282 | 190 | 188
Completed | 265 | 184 | 182
Not Completed | 21 | 7 | 8
Not completed — Decision by Sponsor | 5 | 4 | 2
Not completed — Withdrawal by Subject | 9 | 1 | 4
Not completed — Lost to Follow-up | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg | Total
Number analyzed (Participants) | 286 | 191 | 190 | 667
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (11.3) | 41.4 (11.3) | 42.9 (11.1) | 42.1 (11.3)
Age, Customized [Count of Participants; unit: Participants]
  18 to 64 years | 285 | 191 | 190 | 666
  65 to 74 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 166 | 160 | 552
  Male | 60 | 25 | 30 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 10 | 26
  Not Hispanic or Latino | 277 | 184 | 180 | 641
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 4 | 0 | 8
  Black or African American | 11 | 10 | 6 | 27
  White | 268 | 176 | 184 | 628
  Other | 3 | 1 | 0 | 4
Prior Migraine Prophylactic Medication [Count of Participants; unit: Participants]
  Yes | 218 | 138 | 136 | 492
  No | 68 | 53 | 54 | 175
Prior Migraine Prophylactic Treatment Failure [Count of Participants; unit: Participants]
  Yes | 200 | 127 | 126 | 453
  No | 86 | 64 | 64 | 214
Region [Count of Participants; unit: Participants]
  North America | 135 | 91 | 89 | 315
  Other | 151 | 100 | 101 | 352
Medication Overuse Status [Count of Participants; unit: Participants] — Medication overuse was defined as any of the following criteria being met during the baseline (BL) phase:
  * ≥ 15 days of simple analgesics (> 3 days/week in each week during BL with at least 5 diary days),
  * ≥ 10 days of triptans (> 2 days/week in each week during BL with at least 5 diary days),
  * ≥ 10 days of ergots (> 2 days/week in each week during BL with at least 5 diary days),
  * ≥ 10 days of combination therapy intake of any combination of ergots, triptans, opiates, combination-analgesic medications or simple analgesics (> 2 days/week in each week during BL with at least 5 diary days).
  Participants
    Yes | 117 | 79 | 78 | 274
    No | 169 | 112 | 112 | 393
Monthly Migraine Days [Mean (Standard Deviation); unit: days] — A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine without aura or a migraine with aura.
  Monthly migraine days were calculated as the number of migraine days in the 4-week baseline phase.
  days | 18.22 (4.73) | 17.85 (4.39) | 17.78 (4.72) | 17.99 (4.63)
Disease Duration of Migraine With or Without Aura [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 285 | 191 | 189 | 665
    (all) | 22.21 (12.63) | 20.71 (12.83) | 21.92 (11.80) | 21.70 (12.46)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine with or without aura.
  The change from baseline in monthly migraine days was calculated as the number of migraine days during the last 4 weeks of the 12-week treatment phase - the number of migraine days during the 4-week baseline phase.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week treatment phase
Population: The efficacy analysis set included participants who received at least 1 dose of study drug and completed at least 1 post-baseline monthly eDiary measurement. The number of participants analyzed includes those with observed data at week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: migraine days / month
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg
Number analyzed (Participants) | 267 | 178 | 182
migraine days / month | -4.18 [-4.86 to -3.50] | -6.64 [-7.47 to -5.81] | -6.63 [-7.45 to -5.80]
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg; The primary endpoint was analyzed using a linear mixed effects model including treatment group, baseline value, stratification factors (region and medication overuse status), scheduled visit, and the interaction of treatment group with scheduled visit; Test type: Superiority — A sequential testing procedure, specifically, the hierarchical gate-keeping procedures and Hochberg method, was used to maintain the 2-sided study-wise type I error at 0.05 between the 2 erenumab doses and the primary and secondary endpoints. This comparison was tested at a 2-sided significance level of 0.04; p < 0.001, Generalized linear mixed model; Difference in LS Means = -2.46, 95% CI 2-sided [-3.52 to -1.39]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 140 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — A sequential testing procedure, specifically, the hierarchical gate-keeping procedures and Hochberg method, was used to maintain the 2-sided study-wise type I error at 0.05 between the 2 erenumab doses and the primary and secondary endpoints. This comparison was tested at a 2-sided significance level of 0.01; p < 0.001, Generalized linear mixed model; Difference in LS Means = -2.45, 95% CI 2-sided [-3.51 to -1.38]

2. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction in Monthly Migraine Days From Baseline
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine without aura or a migraine with aura. Monthly migraine days were calculated as the number of migraine days in the 4-week baseline phase and during the last 4 weeks of treatment.
  At least a 50% reduction from baseline in monthly migraine days was determined if the change in monthly migraine days from the 4-week baseline phase to the last 4 weeks of the 12-week treatment phase * 100 / baseline monthly migraine days was less than or equal to -50%.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week treatment phase
Population: The efficacy analysis set included participants who received at least 1 dose of study drug and completed at least 1 post-baseline monthly eDiary measurement.
  Participants with missing post-baseline data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg
Number analyzed (Participants) | 281 | 188 | 187
percentage of participants | 23.5 | 39.9 | 41.2
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg; Analyzed using a Cochran-Mantel-Haenszel test after the missing data were imputed as non-response, stratified by stratification factors (region and medication overuse status); Test type: Superiority — This comparison was tested at a 2-sided significance level of 0.04; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.46 to 3.27]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 140 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — This comparison was tested at a 2-sided significance level of 0.01; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.56 to 3.51]

3. Secondary Outcome: Change From Baseline in Monthly Acute Migraine-specific Medication Treatment Days
Description: Monthly acute migraine-specific medication treatment days is the number of days on which migraine specific medications were used between monthly doses of study drug. Migraine-specific medications includes two categories of medications: triptan-based migraine medications and ergotamine-based migraine medications.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week treatment phase
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: acute migraine treatment days / month
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg
Number analyzed (Participants) | 267 | 178 | 182
acute migraine treatment days / month | -1.58 [-2.05 to -1.11] | -3.45 [-4.02 to -2.87] | -4.13 [-4.70 to -3.56]
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg; Analyzed using a linear mixed effects model including treatment group, baseline value, stratification factors (region and medication overuse status), scheduled visit, and the interaction of treatment group with scheduled visit; Test type: Superiority — This comparison was tested at a 2-sided significance level of 0.04; p < 0.001, Generalized linear mixed model; Difference in LS Means = -1.86, 95% CI 2-sided [-2.60 to -1.13]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 140 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — This comparison was tested at a 2-sided significance level of 0.01; p < 0.001, Generalized linear mixed model; Difference in LS Means = -2.55, 95% CI 2-sided [-3.28 to -1.82]

4. Secondary Outcome: Change From Baseline in Cumulative Monthly Headache Hours
Description: The cumulative duration of any qualified headache between monthly doses of study drug regardless of acute treatment use.
  A qualified headache was defined as follows:
  * a qualified migraine headache (including an aura-only event that is treated with acute migraine-specific medication), or
  * a qualified non-migraine headache, which is a headache that lasted continuously for ≥ 4 hours and was not a qualified migraine headache, or
  * a headache of any duration for which acute headache treatment was administered.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week treatment phase
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: hours / month
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg
Number analyzed (Participants) | 267 | 178 | 182
hours / month | -55.22 [-66.38 to -44.06] | -64.76 [-78.34 to -51.17] | -74.53 [-88.05 to -61.01]
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — This comparison was tested at a 2-sided significance level of 0.04; p = 0.28, Generalized linear mixed model; Difference in LS Means = -9.54, 95% CI 2-sided [-26.98 to 7.90]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 140 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — This comparison was tested at a 2-sided significance level of 0.01; p = 0.030, Generalized linear mixed model; Difference in LS Means = -19.31, 95% CI 2-sided [-36.71 to -1.92]

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4, where:
  Grade 1 = Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2 = Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL); Grade 3 = Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL; Grade 4 = Life-threatening consequences; urgent intervention indicated Grade 5 = Death related to AE.
Time Frame: From the first dose of study drug up to 16 weeks after the last dose (24 weeks)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg
Number analyzed (Participants) | 282 | 190 | 188
Participants
  Any adverse event | 110 | 83 | 88
  AEs grade ≥ 2 | 65 | 45 | 42
  AEs grade ≥ 3 | 13 | 11 | 4
  AEs grade ≥ 4 | 0 | 1 | 0
  Serious adverse events | 7 | 6 | 2
  AEs leading to discontinuation of study drug | 2 | 0 | 2
  Fatal adverse events | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Who Developed Antibodies to Erenumab
Description: Blood samples were first tested in an electrochemiluminescence (ECL)-based bridging immunoassay to detect anti-drug antibodies (ADA) against erenumab. Samples confirmed to be positive for binding antibodies were subsequently tested in a cell-based bioassay to determine neutralizing activity against erenumab (Neutralizing Antibody Assay).
  Developing antibody incidence indicates participants with a negative or no result at baseline and a positive result at any time post-baseline.
  If a sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the sample was defined as positive for neutralizing antibodies.
Time Frame: Baseline and weeks 2, 4, 8, 12 and 24
Population: Randomized participants who received at least one dose of study drug and with available post-baseline antibody data. This endpoint was analyzed in the erenumab treatment groups only.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg
Number analyzed (Participants) | 0 | 189 | 187
Participants
  Binding antibody positive |  | 11 | 3
  Neutralizing antibody positive |  | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 16 weeks after the last dose (a total of 24 weeks)
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Erenumab 70 mg | Erenumab 140 mg
Serious Adverse Events (participants affected / at risk) | 7/282 | 6/190 | 2/188
Other Adverse Events (participants affected / at risk) | 16/282 | 6/190 | 3/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=282) | Erenumab 70 mg (N=190) | Erenumab 140 mg (N=188)
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=282) | Erenumab 70 mg (N=190) | Erenumab 140 mg (N=188)
Nasopharyngitis (Infections and infestations) | 16 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.